CLINICAL TRIAL: NCT04787822
Title: Long Term Follow up of the Lung Transplant Outcomes Group Cohort
Brief Title: Long Term Follow up of the LTOG Cohort
Acronym: LTOG
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Columbia University (Other); University of Alabama at Birmingham (Other); Stanford University (Other); Johns Hopkins University (Other); University of Michigan (Other); University of Pittsburgh (Other); Duke University (Other); Indiana University (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 834898; U01HL145435 (NIH)
Record Dates: First submitted 2021-02-22; First posted 2021-03-09 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Lung Transplant Failure and Rejection
Keywords: Chronic lung allograft dysfunction; Functional status; Lung transplantation
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and buffy coat
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to follow participants who enrolled in the Lung Transplant Outcomes Group. Clinical data, functional assessments, and surveys will be collected to determine long term graft function and functional status of lung transplant recipients.

DETAILED DESCRIPTION:
This project will involve both retrospective and prospective data collection from participants enrolled in the LTOG cohort studies. We will perform long-term Chronic Lung Allograft Dysfunction (CLAD) phenotyping of lung transplant recipients who participated in the LTOG cohort studies utilizing data collected for routine clinical visits. Surviving lung transplant recipients who participated in the LTOG cohort studies will be recruited to enroll in the longitudinal portion of the project. The longitudinal component will include follow-up data collection at 6 month intervals while alive until study termination, study withdrawal, or no longer being seen for follow-up at the participating center. Follow-up data collection will include clinical data collected by study coordinators by reviewing medical records, functional assessment through administration of the Short Physical Performance Battery (SPPB), blood collection and surveys. Data from this project will be linked to data and samples collected during the LTOG cohort or ancillary studies.

ELIGIBILITY:
Inclusion criteria

Long-term phenotyping of CLAD

* Lung transplant recipients who have previously enrolled in the LTOG cohort studies at one of the participating centers

Long-term functional status and well-being

* Lung transplant recipients who have previously enrolled in the LTOG cohort studies at one of the participating centers
* Alive

Exclusion Criteria

Long-term phenotyping of CLAD

* Lung transplant recipient not enrolled in LTOG cohort research studies

Long-term functional status and well-being

* Lung transplant recipient not enrolled in the LTOG cohort research studies
* Lung transplant recipient not receiving post-transplant follow-up care at a participating LTOG center

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Lung transplant recipients who have previously enrolled in the LTOG cohort studies at one of the participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Chronic Lung Allograft Dysfunction (CLAD) phenotyping | From date of transplant to the development of CLAD, up to 25 years
  Change in pulmonary function measured by serial pulmonary function tests (PFTs) and data collected at clinical care visits will be used to assess CLAD.
Functional status phenotyping | From date of transplant to until study termination, withdrawal, or no longer being seen for follow-up at the participating center, up to 25 years
  Change in functional status will be measured by the Short Physical Performance Battery (SPPB). The SPPB is a 3-construct measure that includes gait speed, chair stands, and balance. Each construct is scored from 0 - 4 yielding an aggregate score ranging from 0 - 12. Lower SPPB scores reflect increased frailty.
Well being phenotyping-LT-VLA | From date of transplant to until study termination, withdrawal, or no longer being seen for follow-up at the participating center, up to 25 years
  Change in well being will be measured by patient reported outcomes including the LT-VLA scale. The LT-VLA scale presents a list of activities and asks respondents to rate their difficulty in performing each one on a 4-point scale. A higher score on the LT-VLA indicates more disability.
Well being phenotyping-LT-QOL | From date of transplant to until study termination, withdrawal, or no longer being seen for follow-up at the participating center, up to 25 years
  Change in well being will be measured by patient reported outcomes including the Lung Transplant Quality of Life (LT-QOL) survey. The Lung Transplant Quality of Life (LT-QOL) survey will be used to measure disease specific QOL. The LT-QOL utilizes 5 point scales for all items. The general quality of life scale is scored so that higher scores indicate better QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Christie, MD, Principal Investigator — University of Pennsylvania; Scott Palmer, MD, Principal Investigator — Duke University; Jonathan Singer, MD, Principal Investigator — University of California, San Francisco
Locations (10):
- United States (10):
  - University of Alabama Birmingham, Birmingham, Alabama
  - University of California San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Indiana University, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Columbia University, New York, New York
  - Duke University, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No